CLINICAL TRIAL: NCT06979557
Title: Ambispective Analysis of Patient Reported Outcomes and Visual Acuity in Patients Undergoing a Refractive Lens Exchange With Bilateral Implantation Odyssey Intraocular Lenses
Brief Title: RLE Outcomes With Bilateral Implantation of Odyssey IOLs
Status: Recruiting | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-25-01
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Refractive Lens Exchange

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Odyssey IOL: Bilateral Implantation with the Odyssey IOL
  Interventions: Device: Odyssey IOL

INTERVENTIONS:
Device: Odyssey IOL — Bilateral implantation with the Odyssey IOL

SUMMARY:
This study is a single center, ambispective study of visual outcomes after successful bilateral implantation of the Odyssey IOL. Subjects will be assessed at least 2 months postoperatively at a single visit. Clinical evaluations will include administration of the AIOLIS questionnaire, as well as measurement of visual acuities at distance, intermediate, and near, monocular (right eye) and binocular defocus curve, and refractive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include 40 patients aged 40 years and older who have a measurable Potential Acuity Meter (PAM) of 20/20 electing to undergo bilateral refractive lensectomy surgery with IOL implantation.

Exclusion Criteria:

* Patients with significant ocular comorbidities (e.g., macular degeneration, glaucoma) or prior intraocular surgery will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be aged 40 years and older who underwent bilateral implantation with the Odyssey IOL.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Binocular Photopic Visual Acuity | 2 months posoperatively
  Measured at distance (6m), intermediate at 66cm, and near visual acuity at 40cm and 33cm.
Monocular Photopic Visual Acuity | 2 months posoperatively
  Measured at distance (6m), intermediate at 66cm, and near visual acuity at 40cm and 33cm.
Monocular Defocus Curve (right eye only) | 2 months posoperatively
Binocular Defocus Curve | 2 months posoperatively

SECONDARY OUTCOMES:
Assessment of IntraOcular Lens Implant Symptoms (AIOLIS) Questionnaire | 2 months posoperatively
  The AIOLIS has 37 questions about symptoms, perceptions of general vision, and frequency of wearing glasses or contact lenses. Lower scores for the symptom questions indicate lower frequency and both of visual disturbances.

OTHER OUTCOMES:
Percentage of patients within ± 0.5 D MRSE | 2 months posoperatively
  Manifest refraction spherical equivalent (MRSE)
Percentage of eyes requiring additional corneal refractive procedures | 2 months postoperative
Correlation between pupil size and defocus curve | 2 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Brunson, OD, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No